CLINICAL TRIAL: NCT00495170
Title: Phase II Concurrent Proton and Chemotherapy in Locally Advanced Stage IIIA/B Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Concurrent Proton and Chemotherapy in Locally Advanced Stage IIIA/B Non-Small Cell Lung Cancer (NSCLC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2004-0976; NCI-2012-01504 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2007-06-28; First posted 2007-07-02 (Estimated); Results first posted 2019-02-06 (Actual); Last update posted 2019-02-06 (Actual); Status verified 2019-01

CONDITIONS: Lung Cancer
Keywords: Non-Small Cell Lung Cancer; Lung Cancer; Proton Radiotherapy; Proton Beam; Paclitaxel; Taxol; Carboplatin; Paraplatin; NSCLC
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Carboplatin; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Concurrent proton and Chemotherapy (Experimental): Proton Radiotherapy + Carboplatin + Paclitaxel
  Interventions: Drug: Carboplatin; Radiation: Proton Radiotherapy; Drug: Paclitaxel

INTERVENTIONS:
Drug: Carboplatin — 2 area under curve (AUC) by vein Weekly
  Other Names: paraplatin
Radiation: Proton Radiotherapy — 2 GY/fraction for 37 fractions (daily treatment, Monday to Friday, for 7.5 weeks).
Drug: Paclitaxel — 50 mg/m^2 by vein Weekly
  Other Names: Taxol

SUMMARY:
The goal of this clinical research study is to learn if proton radiotherapy given with standard chemotherapy (such as paclitaxel and carboplatin) can help to control locally advanced NSCLC. The safety of this treatment will also be studied.

DETAILED DESCRIPTION:
A proton beam is made up of charged particles that have a well-defined range of penetration into tissues. How deep it can penetrate is decided by both the beam's energy and the density of the tissue through which it passes. As the proton beam penetrates the body, the particles slow down, and the beam deposits its dose sharply near the end of its range. This is a phenomenon known as the Bragg peak. By adjusting the Bragg peak, the doctor can deliver a full, localized, uniform dose of energy to the treatment site while sparing the surrounding normal tissues. The proton beam is ideal for treatments where organ preservation is very important, such as lung cancer.

If you are found to be eligible to take part in this study, you will receive 37 treatments of proton radiotherapy (Monday through Friday for 7 1/2 weeks). During the treatment, you will lie still on a table for about 30-45 minutes per day in the same position. The proton machine will deliver the dose according to the plan designed by the physician and controlled by a computer. You will not feel, see, or smell anything during the proton beam delivery. While on study, you will also be receiving weekly standard low-dose chemotherapy possibly followed by full-dose chemotherapy.

During the treatment, you will be seen by a doctor and research nurse once a week to evaluate possible side effects. You will have a physical exam and you will have a medical history. About 2 teaspoons of blood will be drawn for routine tests.

You will be taken off study early if the disease gets worse or intolerable side effects occur. After finishing the treatment, 6 week follow up is recommended after completion of radiotherapy, then required every 3 months (+1 month) for 2 years, then every 6 months (+1 month) for 3 years, and then once a year for 2 years. You will have imaging tests (chest CT or positron emission computed tomography (PET) scan) and routine blood tests (about 2 teaspoons) at the follow-up visits.

This is an investigational study. Proton radiotherapy is FDA approved for the treatment of lung cancer. A total of 65 patients will be take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically documented NSCLC.
2. Inoperable stage IIIA (T1--3N2MO, T3N1MO) and IIIB (T1-3N3MO, T4NO-3MO) disease excluding malignant pleural effusion.
3. Performance score Karnofsky Performance Status (KPS) 70-100, Weight loss: less or equal to 10% in 6 months prior to diagnosis.
4. Patient consented for the protocol
5. Induction chemotherapy is allowed.

Exclusion Criteria:

1. Prior chest radiotherapy.
2. Previous or concomitant malignancy other than (a) curatively treated carcinoma in situ of cervix, (b) basal cell carcinoma of the skin, (c) curatively treated superficial transitional cell carcinoma of the urinary bladder, and (d) early stage tumor treated more than 3 years ago for cure.
3. Pregnancy. Patients (men and women) of child bearing potential should use an effective (for them) method of birth control throughout their participation in this study.
4. Off study criteria: a) If a patient is found to have distant metastasis during treatment and/or immediate after the treatment (<60 days) indicating inaccurate cancer stage, he or she will be taken off study. b) If a patient does not follow up at MD Anderson and does not forward his or her medical records such as CT, PET/CT, pulmonary function test (PFT) or pathology report as required by protocol, he or she will be taken off study. c) If a patient does not have any required post-treatment evaluation such as images, he or she will be taken off study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2006-04-14 (Actual); Primary Completion 2017-06-14 (Actual); Study Completion 2017-06-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joe Y. Chang, MD, PhD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Koay EJ, Lege D, Mohan R, Komaki R, Cox JD, Chang JY. Adaptive/nonadaptive proton radiation planning and outcomes in a phase II trial for locally advanced non-small cell lung cancer. Int J Radiat Oncol Biol Phys. 2012 Dec 1;84(5):1093-100. doi: 10.1016/j.ijrobp.2012.02.041. Epub 2012 Apr 27. PMID 22543217
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Inoperable stage III NSCLC with KPS of 70-100, medically fit to receive concurrent and/or induction chemotherapy, weight loss ≤ 10% in the 6 months before diagnosis, provide informed consent. Patients were not enrolled in cases of prior chest radiation therapy and/or pregnancy, with prior and/or concomitant malignant neoplasms.
Groups:
- Concurrent Proton and Chemotherapy: Weekly infusions of carboplatin (area under the curve of 2 units) and paclitaxel (50mg/m2) with concurrent passively scattered PBT (74-Gy relative biological effectiveness)
Period: Overall Study
Arm/Group | Concurrent Proton and Chemotherapy
Started | 84
Completed | 64
Not Completed | 20
Not completed — Lost to Follow-up | 9
Not completed — Withdrawal by Subject | 3
Not completed — Inappropriate staging | 8

BASELINE CHARACTERISTICS:
Population: There were 64 out of 84 patients treated under the protocol and evaluable for data analysis.
Arm/Group | Concurrent Proton and Chemotherapy
Number analyzed (Participants) | 64
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 44
Age, Continuous [Median (Full Range); unit: years] | 70 [37 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 42
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 60
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants] — Population: There were 64 out of 84 patients treated under the protocol and evaluable for data analysis.
  Participants
    United States | 63
    Bahamas: number analyzed (Participants) | 1
    Bahamas | 1
Non-small cell lung cancer (NSCLC) histological Subtype [Count of Participants; unit: Participants]
  Squamous cell carcinoma | 28
  Adenocarcinoma | 25
  Non-small cell lung cancer, not otherwise specific | 11
Patients with Stage III Non-Small Cell Lung Cancer Gross tumor volume [Median (Full Range); unit: cm^3] | 87 [4.1 to 753.2]
Patients with Stage III Non-Small Cell Lung Cancer Karnofsky performance status at diagnosis [Median (Full Range); unit: units on a scale] — Population: The Karnofsky Performance Score (KPS) ranking runs from 100 to 0, where 100 is "perfect" Normal health and 0 is death. Practitioners occasionally assign performance scores in between standard intervals of 10. The KPS was to allow physicians to evaluate a patient's survival.
  The higher KPS scores, the better treatment outcome.
  units on a scale | 90 [70 to 100]
American Joint Committee on Cancer (AJCC) disease staging [Count of Participants; unit: Participants] — AJCC-TNM staging(6th): IIIA:T(1-3)N2M0;T3N1M0;IIIB:T(1-3)N3M0;T0:No evidence of primary tumor;T1:Tumor≤3cm;T2:tumor>3cm;involve:main bronchus,visceral pleura or≥2cm to Carina;atelectasis or pneumonia;T3:Invades:chestwall,diaphragm,mediastinal pleura,parietal pericardium,or tumor<2cm to Carina,entire lung atelectasis or pneumonia;T4 invades:mediastinum,heart,great vessels,separate tumor.N0:No regional LN;N1:ipsilateral peribroncheal and/or hilar LN;N2:ipsilateral mediastinal and/or subcrinal LN;N3:contralateral mediastinal,hilar LN;scalence or supraclavicalar LN;Earlier staging,better outcome.
  Participants
    Stage IIIA | 30
    Stage IIIB | 34
American Joint Committee on Cancer (AJCC) TNM Categories - Primary Tumor [Count of Participants; unit: Participants] — AJCC-TNM staging(6th): T0:No evidence of primary tumor; T1:Tumor≤3cm; T2:tumor>3cm;involve:main bronchus,visceral pleura or≥2cm to Carina;atelectasis or pneumonia; T3:Invades:chestwall,diaphragm,mediastinal pleura,parietal pericardium,or tumor<2cm to Carina,entire lung atelectasis or pneumonia;T4 invades:mediastinum,heart,great vessels,separate tumor.
  Participants
    T0-2 | 37
    T3-4 | 27
American Joint Committee on Cancer (AJCC) TNM Categories - Lymph Nodes [Count of Participants; unit: Participants] — AJCC-TNM staging(6th): N0:No regional LN;N1:ipsilateral peribroncheal and/or hilar LN;N2:ipsilateral mediastinal and/or subcrinal LN;N3:contralateral mediastinal,hilar LN;scalence or supraclavicalar LN;Earlier staging,better outcome.
  Participants
    N0-1 | 6
    N2-3 | 58
Patients with Stage III Non-Small Cell Lung Cancer Chemotherapy Types [Count of Participants; unit: Participants] — Population: Patients will receive the weekly carboplatin and paclitaxel concurrent chemotherapy. Additional "consolidation" or adjuvant chemotherapy may be given >/= 4 weeks after concurrent chemo/RT at the discretion of the treating medical oncologist based upon the patient's performance status and recovery from toxicities of the concurrent chemo/RT.
  Participants
    Induction | 20
    Concurrent | 64
    Adjuvant | 18
Patients with Stage III Non-Small Cell Lung Chemotherapy Cycles [Median (Full Range); unit: cycles]
  Chemotherapy Induction Cycle | 2 [1 to 6]
  Chemotherapy Concurrent Cycle | 7 [3 to 8]
  Chemotherapy Adjuvant Cycle | 8 [1 to 8]

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival and Progression Free Survival
Description: The primary objective was to improve overall survival (OS). Patients are recommended to have follow up 6 weeks after completion of concurrent chemo radiotherapy for the evaluation of acute treatment toxicities, then required every 3 months (+ 1 month) for two years, then every 6 months (+ 1 month) for three years and then annually for the rest of their lives, that is standard of care.
  Statistics were performed with Strata/MP 14.2 software. OS was calculated by Kaplan-Meier Methodology (K-M) from the beginning of enrollment to date of death or last follow-up.
  Progression-free survival (PFS) was defined from enrollment to any treatment failure or death. PFS will be evaluated by series CT of chest with contrast for every follow up except 6 weeks after the concurrent chemo radiotherapy for two years.
  Multivariate Cox proportional hazards modeling was used to examine predictors of OS when adjusting for each of the collected potential confounding variables.
Time Frame: The Overall survival (OS): From date of registration to the last follow-up (f/u), or lost to f/u, or death up to 5 years. The progression free survival (PFS): From date of registration to the date of first documented progression or death up to 5 years.
Population: Kaplan-Meier analysis of overall survival (OS), progression-free survival (PFS), actuarial distant metastasis, and local regional recurrence. Patterns of treatment failure were categorized as local/regional or distant. Acute and late toxic effects were prospectively assigned using Common Terminology Criteria for Adverse Events, v3.0.
Measure: Number; unit: percentage of participants
Arm/Group | Concurrent Proton and Chemotherapy
Number analyzed (Participants) | 64
percentage of participants
  Overall Survival at 5 years | 29
  Progression Free Survival (PFS) | 12.9
  Progression Free Survival at 5 years | 22

ADVERSE EVENTS:
Time Frame: From the time of registration to the adverse event start date, assessed up to 5 years.
Description: During treatment, acute radiation adverse events will be evaluated weekly according to National Cancer Institute Common Toxicity Criteria version 3. Only grade ≥2 toxicity directly related to therapy will be documented. Pre-treatment symptoms is not required to be documented except it gets worse.
  Post-treatment:
  Patients are follow up 6 weeks after completion of concurrent chemoradiotherapy, then every 3 months for 2 years, every 6 months for 3 years.
Arm/Group | Concurrent Proton and Chemotherapy
All-Cause Mortality (participants affected / at risk) | 47/64
Serious Adverse Events (participants affected / at risk) | 35/64
Other Adverse Events (participants affected / at risk) | 0/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Concurrent Proton and Chemotherapy (N=64)
Lobar atelectasis (Respiratory, thoracic and mediastinal disorders) | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 7
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 0
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 8
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0
Constipation (Gastrointestinal disorders) | 0
Diarrhea (Gastrointestinal disorders) | 0
Dyspepsia (Gastrointestinal disorders) | 0
Dysphagia (Gastrointestinal disorders) | 0
Esophagitis (Gastrointestinal disorders) | 7
Esophageal stricture (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 0
Nausea (Gastrointestinal disorders) | 1 (11)
Odynophagia (Gastrointestinal disorders) | 0
Vomiting (Gastrointestinal disorders) | 0
Arrhythmia (Cardiac disorders) | 0
Palpitations (Cardiac disorders) | 0 (0)
Tachycardia (Cardiac disorders) | 0
Uremia (Metabolism and nutrition disorders) | 0 (0)
Blood urea nitrogen increase (Metabolism and nutrition disorders) | 0
Elevated creatinine (Metabolism and nutrition disorders) | 0
Anemia (Metabolism and nutrition disorders) | 4 (35)
Hypocalcemia (Metabolism and nutrition disorders) | 0
Hypomagnesemia (Metabolism and nutrition disorders) | 0
Hyponatremia (Metabolism and nutrition disorders) | 3
Hypotension (Metabolism and nutrition disorders) | 1 (1)
Leukopenia (Metabolism and nutrition disorders) | 15 (57)
Lymphopenia (Metabolism and nutrition disorders) | 0
Neutropenia (Metabolism and nutrition disorders) | 3
Thrombocytopenia (Metabolism and nutrition disorders) | 0
Anorexia (General disorders) | 0
Dehydration (General disorders) | 4
Dermatitis (General disorders) | 6
Dizziness (General disorders) | 0
Fatigue (General disorders) | 7
Fever (General disorders) | 2
Hyperpigmentation (General disorders) | 0
Pain (General disorders) | 2
Pruritus (General disorders) | 1
Rash (General disorders) | 1
Sourness (General disorders) | 0
Weight loss (General disorders) | 4
Alopecia (Skin and subcutaneous tissue disorders) | 0
Anxiety (Psychiatric disorders) | 0
Candidiasis (Skin and subcutaneous tissue disorders) | 1
Infection (Infections and infestations) | 1
Insomnia (Social circumstances) | 0
Muscle weakness (Musculoskeletal and connective tissue disorders) | 0
Peripheral motor neuropathy (Nervous system disorders) | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0
Lung atelectasis (Respiratory, thoracic and mediastinal disorders) | 0
Dysphagia (Respiratory, thoracic and mediastinal disorders) | 0
Bronchial fistula (Respiratory, thoracic and mediastinal disorders) | 1
Bronchial stricture (Respiratory, thoracic and mediastinal disorders) | 0
Pericardial effusion (Cardiac disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2010-12-06): https://cdn.clinicaltrials.gov/large-docs/70/NCT00495170/Prot_SAP_000.pdf